CLINICAL TRIAL: NCT06520618
Title: Clinical Study on the Efficacy and Safety of Qingre Heji in the Treatment of Acute Upper Respiratory Tract Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Li Naijing, Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M1112
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Acute Upper Respiratory Tract Infection; Traditional Chinese Medicine; Randomised Controlled Trial

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Drug: Qing Re He Ji
- Control Group (Active Comparator)
  Interventions: Drug: Shuanghuanglian Oral Liquid

INTERVENTIONS:
Drug: Qing Re He Ji — Oral administration of Qing Re He Ji
  Arms: Experimental Group
Drug: Shuanghuanglian Oral Liquid — Oral administration of Shuanghuanglian Oral Liquid
  Arms: Control Group

SUMMARY:
Originating from China, TCM complements conventional approaches by alleviating symptoms, balancing physical conditions, and enhancing immunity. Clinical studies have shown TCM to be safe and effective in treating AURI. In TCM syndrome differentiation, AURI is considered a "Wind-Heat Syndrome", requiring treatment that clears heat and detoxifies the body. Qing Re He Ji (QRHJ; heat-clearing mixture), a TCM compound developed by our hospital, comprises Huang Qin (Radix Scutellariae), Da Qing Ye (Folium Isatidis), Ge Gen (Radix Puerariae), Yin Chen (Herba Artemisiae Scopariae), and Guan Zhong (Cyrtomium Rhizome). Widely used for AURI, QRHJ effectively clears heat, eliminates pathogens, and strengthens healthy qi. Clinical applications have demonstrated its efficacy, complemented by significant advancements in animal experiments and pharmacokinetics research. To further validate these results, systematic clinical research is imperative, especially in the context of limited direct comparisons between QRHJ and other commercially available TCMs like Shuang Huang Lian (SHL) oral liquid, known for its efficacy and safety in AURI treatment.

Therefore, we performed a rigorously designed non-inferiority randomised controlled trial to assess the efficacy and safety of QRHJ in treating AURI in adults, comparing it directly with SHL oral liquid. This study aimed to bridge existing research gaps and provide healthcare professionals with more diversified treatment options, thereby enhancing personalised and comprehensive patient care plans. Furthermore, we hope that our findings will establish a scientific basis for integrating TCM into modern healthcare practices, promoting the synergy of Chinese and Western medicine.

ELIGIBILITY:
Inclusion Criteria:

* 1: Voluntarily sign informed consent

  2: Age ≥ 18 years old

  3: Meet the diagnostic criteria of acute respiratory tract infection: Internal Medicine edited by chenhaozhu (9th Edition, people's Health Publishing House)

Exclusion Criteria:

* 1: Legal infectious diseases with upper respiratory symptoms

  2: Patients with severe pneumonia

  3: Severe primary diseases such as cardiovascular, cerebrovascular, liver, kidney and hematopoietic system

  4: After this episode, he has received other antiviral, anti-inflammatory, antipyretic and analgesic drugs or any other drugs to treat colds

  5: Pregnant or lactating women

  6: Allergic constitution and drug allergy

  7: Psychopath

  8: Those who have participated in other clinical trials within three months

  9: Persons with a history of drug abuse

  10: Other circumstances that the investigator believes are not suitable for enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Overall Symptom and Sign Score Improvement Rate | At days 0 (baseline) and 6
  We use both traditional Chinese medicine (TCM) and Western medicine scales to assess the condition.
Onset time | At days 0 (baseline) and 6
  Defined as the duration from medication administration to a 0.5°C decrease in body temperature.
Antipyretic time | At days 0 (baseline) and 6
  Measured as the time taken for axillary temperature to drop below 37.3°C after the first dose and maintained for at least 24 hours without recurrence
Single Symptom and Sign Disappearance Rate | At days 0 (baseline) and 6
  Disappearance rate of individual TCM symptoms and signs

CONTACTS AND LOCATIONS:
Overall Officials: Difei Wang, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No
One years after the article was published, disclose the original data if necessary.